CLINICAL TRIAL: NCT06903819
Title: Ketamine's Impact on Opioid Use, Pain, and Mental Health in Polytraumatized Orthopedic Patients: A Randomized Controlled Trial (KOPM)
Brief Title: Ketamine for Pain, Opioid Use, and Mental Health in Orthopedic Trauma Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2025-75
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Orthopedic Trauma Surgery Patients; Postoperative Pain; Opioid Use; Depression; Post-traumatic Stress Disorder (PTSD)
Keywords: Ketamine; Orthopedic Trauma; Postoperative Pain; Opioid Reduction; Depression; PTSD; Musculoskeletal Injury; Trauma Surgery
MeSH Terms: conditions — Pain, Postoperative; Depression; Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Masking Description: Participants are blinded to group assignment. The anesthesia team is unblinded to ensure safe intraoperative management. Postoperative clinical teams and study personnel conducting follow-up assessments remain blinded. An unblinding log will document any instances where treatment assignment becomes known.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Experimental): Participants in this group will receive a single intraoperative dose of intravenous (IV) ketamine (0.5 mg/kg) within 30 minutes of anesthesia induction. The intervention is designed to assess ketamine's effects on postoperative pain, opioid use, and symptoms of depression and PTSD in patients undergoing surgical fixation for musculoskeletal trauma.
  Interventions: Drug: Ketamine
- Control Group (Active Comparator): Participants in this group will receive standard general anesthesia without ketamine. This group serves as a comparison to evaluate the effectiveness of ketamine on postoperative pain levels, opioid consumption, and psychological recovery following orthopedic trauma surgery.
  Interventions: Drug: standard general anesthesia

INTERVENTIONS:
Drug: Ketamine — Participants in this group will receive a single intravenous (IV) dose of ketamine at 0.5 mg/kg, administered within 30 minutes of anesthesia induction during surgical fixation for musculoskeletal trauma. The purpose of the intervention is to evaluate ketamine's effect on postoperative pain, opioid consumption, and psychological recovery, including symptoms of depression and post-traumatic stress disorder (PTSD).
  Arms: Ketamine Group
Drug: standard general anesthesia — Participants in this group will receive standard general anesthesia during surgical fixation for musculoskeletal trauma. No ketamine will be administered. This group serves as a comparison to evaluate the effects of ketamine on pain, opioid use, and psychological recovery.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if ketamine, given during surgery, can help improve recovery for adults with serious orthopedic trauma. The study will test whether ketamine reduces pain, lowers the need for opioids, and improves mental health outcomes like depression and post-traumatic stress disorder (PTSD).

The main questions it aims to answer are:

Does ketamine reduce pain after surgery compared to standard anesthesia?

Does ketamine reduce the amount of opioids patients need for pain control?

Does ketamine improve symptoms of depression and PTSD after orthopedic trauma?

Researchers will compare patients who receive ketamine during surgery with those who receive standard anesthesia without ketamine to see if ketamine helps improve both physical and psychological recovery.

Participants will:

Be randomly assigned to receive either a single dose of ketamine or standard anesthesia during surgery.

Report their pain using a simple pain scale (Visual Analog Scale, VAS).

Complete short surveys about mood and mental health (PHQ-9 for depression and PCL-5 for PTSD) at several time points after surgery.

Allow the research team to review their electronic medical records to measure opioid prescriptions during recovery.

Attend follow-up visits in clinic or by secure telehealth (e.g., Zoom) at 1-7 days, 2-3 weeks, 6 weeks, 3 months, and 6 months after surgery

DETAILED DESCRIPTION:
Orthopedic trauma patients often face challenges in both physical and psychological recovery following injury. Pain control is difficult, as effective pain relief must be balanced against the risks of opioid dependence. In addition, rates of depression and post-traumatic stress disorder (PTSD) are high in this population, further complicating recovery. These overlapping challenges highlight the need for new approaches that address both pain and mental health outcomes.

Ketamine, a commonly used anesthetic, has properties that may benefit trauma patients beyond its routine role in surgery. Evidence suggests that low-dose intravenous (IV) ketamine can reduce acute postoperative pain, decrease the need for opioid medications, and have rapid effects on depressive symptoms. Some studies also indicate that ketamine may reduce PTSD-related symptoms by influencing brain pathways involved in stress and memory. However, despite these promising effects, ketamine has not been fully integrated into trauma care protocols, in part due to limited large-scale data in orthopedic populations.

This single-blind randomized controlled trial is designed to evaluate whether a single intraoperative dose of IV ketamine (0.5 mg/kg) improves recovery in adults undergoing surgical fixation for musculoskeletal trauma. Participants will be randomly assigned to receive either ketamine or standard anesthesia without ketamine. While the anesthesia team will be aware of group assignment to ensure patient safety, participants and postoperative care teams will remain blinded.

The study will measure multiple aspects of recovery, including:

Postoperative pain intensity, using a validated Visual Analog Scale (VAS).

Opioid consumption during recovery, quantified from electronic medical records and converted to morphine milligram equivalents (MME).

Psychological outcomes, including symptoms of depression and PTSD, assessed with the PHQ-9 and PCL-5 surveys at defined follow-up intervals.

Follow-up assessments will occur at several time points after surgery, ranging from the early postoperative period (1-7 days) to longer-term recovery (up to 6 months). To accommodate patients unable to attend in-person visits, telehealth-based follow-up is available.

By focusing on both physical and psychological outcomes, this trial aims to determine whether ketamine can serve as a dual-purpose intervention in orthopedic trauma care. Results will provide evidence on the feasibility and potential benefits of incorporating ketamine into standard surgical practice for patients with severe musculoskeletal injuries.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65
* Undergoing acute operative fixation for musculoskeletal trauma
* Injury Severity Score (ISS) greater than 15
* Ability to provide informed consent (or consent provided by a legally authorized representative)

Exclusion Criteria:

* Age under 18 or over 65
* Use of ketamine for preoperative or postoperative sedation
* Known allergy or contraindication to ketamine
* Prior unsuccessful ketamine therapy for major depressive disorder (MDD) or PTSD
* Severe psychiatric conditions or psychotic features
* History of dementia or glaucoma
* Currently engaged in trauma-focused cognitive behavioral therapy or PTSD psychotherapy started within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (VAS) | 1-7 days, 2-3 weeks (±1 week), 6 weeks (±2 weeks), 3 months (±3 weeks), and 6 months (±5 weeks) postoperatively.
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a validated 0-100 continuous scale (or 0-10 categorical equivalent). Higher scores indicate greater pain. This outcome evaluates whether intraoperative ketamine reduces postoperative pain compared to standard anesthesia.

SECONDARY OUTCOMES:
Postoperative Opioid Consumption (MME) | 1-7 days, 2-3 weeks (±1 week), 6 weeks (±2 weeks), 3 months (±3 weeks), and 6 months (±5 weeks) postoperatively.
  Opioid use will be quantified from prescription records in the electronic medical record (EMR) and converted into morphine milligram equivalents (MME). This will assess whether intraoperative ketamine reduces opioid requirements compared to the control group.

OTHER OUTCOMES:
Depression Symptoms (PHQ-9) | 1-7 days, 2-3 weeks (±1 week), 6 weeks (±2 weeks), 3 months (±3 weeks), and 6 months (±5 weeks) postoperatively.
  Depression severity will be measured with the Patient Health Questionnaire-9 (PHQ-9), a validated self-report survey. Higher scores indicate greater depressive symptom burden.
PTSD Symptoms (PCL-5) | 1-7 days, 2-3 weeks (±1 week), 6 weeks (±2 weeks), 3 months (±3 weeks), and 6 months (±5 weeks) postoperatively.
  Post-traumatic stress disorder symptoms will be measured using the PTSD Checklist for DSM-5 (PCL-5), a validated self-report survey. Higher scores indicate more severe PTSD symptoms.
Adverse Events Related to Ketamine | Monitored continuously through 6 months postoperatively.
  Frequency and severity of adverse events (e.g., nausea, vomiting, dizziness, hypertension, dissociative symptoms, allergic reactions, or prolonged psychotomimetic effects) will be recorded. Participants scoring ≥20 on the PHQ-9 or ≥50 on the PCL-5 will trigger automated alerts and referral to psychiatric care. All serious adverse events (SAEs) related or possibly related to ketamine will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Max Evan Davis, MD, Principal Investigator — Texas Tech University Health Sciences Center Department of Orthopaedic Surgery,
Locations (2):
- United States (2):
  - Texas Tech University Health Sciences Center Lubbock, Lubbock, Texas
  - University Medical Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No
Only aggregate results will be published or shared in accordance with ethical guidelines.